CLINICAL TRIAL: NCT01850862
Title: Progressive Collective-exercise Program on the Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Wouber Hérickson de Brito Vieira, PhD, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP-UFRN 530/11
Record Dates: First submitted 2013-05-04; First posted 2013-05-10 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Collective group exercise program in patients with KOA (Experimental): Collective exercises program for patients with osteoarthritis and orientation about this disease
  Interventions: Other: Collective group exercise program in patients with KOA
- Control group (without exercise) (Active Comparator): Orientation about osteoarthritis disease but without any exercise program
  Interventions: Other: Orientation (without exercise)

INTERVENTIONS:
Other: Collective group exercise program in patients with KOA
  Arms: Collective group exercise program in patients with KOA
Other: Orientation (without exercise) — Orientation about osteoarthritis disease but without any exercise program
  Arms: Control group (without exercise)

SUMMARY:
The investigators hypothesized that an eight-week collective group exercise program would improve pain, quality of life and functional capacity in patients with knee osteoarthritis (KOA) compared with those receiving no exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic and moderate to severe medical diagnostic of KOA.
* Subjects with normal cognitive functions and no restriction to perform physical activities were recruited from the hospital's KOA database and eligible to participate if they had presented: Lequesne questionnaire criteria (5 - 13.5), knee pain score between 3 and 7 (on a 0 -10 Visual Analogue Scale), stable doses of non-steroidal anti-inflammatory drugs (NSAIDs) and no regular physical exercise or use of canes in the months prior to the study.

Exclusion Criteria:

* Symptomatic heart disease; symptomatic disease of the lower limbs (other than KOA); symptomatic lung disease; severe systemic disease; severe psychiatric illness; regular physical exercise (three or more times per week for at least 3 months); drug injection in the knee in the previous 3 months; physiotherapy on the lower limbs in the previous 3 months and absence in two consecutive training sessions or three nonconsecutive sessions

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Pain | Eight weeks
  pain assessed by Visual Analogue Scale

SECONDARY OUTCOMES:
quality of life | Eight weeks
  quality of life assessed by SF-36 questionnaire

OTHER OUTCOMES:
functional capacity | Eight weeks
  functional capacity assessed by Lequesne questionnaire and functional tests.

CONTACTS AND LOCATIONS:
Overall Officials: Wouber Hérickson de Brito Vieira, PhD, Principal Investigator — Universidade Federal do Rio Grande do Norte; Bento João Abreu, PhD, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (1):
- Federal University of Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil

REFERENCES:
- [Derived] da Silva FS, de Melo FE, do Amaral MM, Caldas VV, Pinheiro IL, Abreu BJ, Vieira WH. Efficacy of simple integrated group rehabilitation program for patients with knee osteoarthritis: Single-blind randomized controlled trial. J Rehabil Res Dev. 2015;52(3):309-22. doi: 10.1682/JRRD.2014.08.0199. PMID 26237073